## STUDY DOCUMENT

Official Study Title:

The Effect of Prone Position on Oxygen Saturation, Blood Gas Parameters, and Respiratory Rate in Intensive Care Patients with COVID-19-induced ARDS

NCT Number: NCTXXXXXXX

Document Type: Informed Consent Form

Document Date: 26 May 2025

Last Updated/Approved: 26 May 2025

### INFORMED CONSENT FORM

# 1. Study Title

The Effect of Prone Position on Oxygen Saturation, Blood Gas Parameters, and Respiratory Rate in Intensive Care Patients with COVID-19-induced ARDS

### 2. Introduction

You are being invited to participate in a research study. Please read this form carefully and ask any questions you may have before agreeing to take part.

# 3. Purpose of the Study

This study aims to investigate whether a short-term prone position can improve oxygen levels and respiratory function in patients with COVID-19-induced ARDS.

#### 4. Procedures

If you agree to participate, you will be randomly assigned to a group. If in the intervention group, you will be placed in a prone position for 30 minutes on two consecutive days. Blood gas levels, oxygen saturation, and respiratory rate will be measured.

# **5. Voluntary Participation**

Your participation in this study is entirely voluntary. You may withdraw at any time without affecting your medical care.

## 6. Risks and Discomforts

The prone position may cause mild discomfort, including pressure-related discomfort in some areas of the body. All necessary precautions will be taken to minimize risk.

#### 7. Benefits

You may experience improved oxygenation. The information gained from this study may help other patients in the future.

## 8. Confidentiality

Your information will be kept confidential. Your name will not appear in any published results. Data will be stored securely and used only for research purposes.

#### 9. Contacts

If you have any questions about this study, please contact:

Dr. Veysel Tekin at veyseltekin571453@gmail.com

### **10. Consent Statement**

I have read and understood the information provided above. I have had the opportunity to ask questions and all of my questions have been answered. I voluntarily agree to participate in this study.

| Participant Name: | |
|------------------------|-------|
| Participant Signature: | Date: |
| Researcher Name: | |
| Researcher Signature: | Date: |